CLINICAL TRIAL: NCT01330121
Title: Pharmacist Discharge Counseling: Bridging the Gap by Transitional Care
Brief Title: Bridging the Gap by Transitional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Leon Fogelfeld MD, Chair, Division of Endocrinology, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB #10-165
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Adherence with discharge diabetes medications; Diabeted mellitus type 2 greater than one year; Patient with provider and prescriptions filled within CCHS
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist Counseling (Active Comparator): Pharmacist Counseling includes but is not limited to:
  Reviewing and explaining their medications (dosing, side effects, route) Reviewing symptoms and complications of hyper and hypoglycemia Defining glycemic & non-glycemic goal levels Explaining the importance of compliance with medications & appointments Educating on the basics of nutrition and physical activity
  Interventions: Other: Pharmacist Counseling
- Standard therapy (No Intervention): Standard therapy: Nurses distribute a education pamphlet on diabetes

INTERVENTIONS:
Other: Pharmacist Counseling — Pharmacist Counseling includes but is not limited to:
  Reviewing and explaining their medications (dosing, side effects, route) Reviewing symptoms and complications of hyper and hypoglycemia Defining glycemic & non-glycemic goal levels Explaining the importance of compliance with medications & appointments Educating on the basics of nutrition and physical activity
  Arms: Pharmacist Counseling

SUMMARY:
The purpose of the study is to evaluate patient adherence with discharge diabetes medications up to 120 days following pharmacist counseling during hospital stay about diabetes self management

DETAILED DESCRIPTION:
It is a prospective, randomized, controlled Study. Patients randomized in a 1:1 ratio to pharmacist counseling or standard of therapy prior to discharge.

Standard therapy: Nurses distribute a education pamphlet on diabetes.

Pharmacist Counseling includes but is not limited to:

* Reviewing and explaining their medications (dosing, side effects, route)
* Reviewing symptoms and complications of hyper and hypoglycemia
* Defining glycemic & non-glycemic goal levels
* Explaining the importance of compliance with medications & appointments
* Educating on the basics of nutrition and physical activity

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18 to 85 years of age
* Historical diagnosis of type 2 diabetes mellitus greater than one year
* HbA1c concentration ≥ 8%
* Discharged from general medicine unit of John H. Stroger Jr, Hospital of Cook County
* Patient with provider and prescriptions filled within CCHS

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnancy
* Major illness or debility, that prohibits the subject from participating in the study
* History of any hemoglobinopathy that may affect determination of HbA1c
* Non-English speaking patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Adherence with discharge diabetes medications up to 120 days following pharmacist counseling during hospital stay about diabetes self management | up to 120 days
  The primary efficacy endpoint will be the difference in rate of adherence with medications Adherence will be assessed at 30, 60, 90, and 120 days following discharge An average of the total adherence rate 120 days following discharge will be calculated as the primary outcome measure

SECONDARY OUTCOMES:
Change in A1c after 90 days | up to 90 days
  A1c measure as % and lipid panel 90 days following pharmacist counseling
  * To demonstrate an improvement in health literacy following pharmacist counseling on diabetes
  * To evaluate patient compliance with follow up appointments up to 90 days following pharmacist counseling
Change in BP after 90 days | up to 90 days
  BP in mm/Hg
Change in lipids after 90 days | up to 90 days
  Lipid measurements in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Leon Fogelfeld, M.D., Principal Investigator — John H. Stroger Hospital of Cook County, Division of Endocrinology; Mansi Shah, PharmD, Principal Investigator — John H. Stroger Hospital of Cook County, Department of Pharmacy; CaTanya Norwood, R.PH, Principal Investigator — John H. Stroger Hospital of Cook County, Department of Pharmacy
Locations (1):
- John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois, United States